CLINICAL TRIAL: NCT00572065
Title: Prospective Pilot Trial of Arsenic Trioxide (Trisenox®) in Combination With Cytosine Arabinoside in Patients With Advanced or Transformed Myelofibrosis
Brief Title: Pilot Trial of Arsenic + Cytarabine in Patients With Myelofibrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0707009291
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Arsenic Trioxide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Experimental): Arsenic trioxide [TrisenoxTM Injection], will be administered at a dose of 0.25 mg/kg on days 1-5 and days 8-12.
  Interventions: Drug: arsenic trioxide; Drug: cytarabine

INTERVENTIONS:
Drug: arsenic trioxide — Cytarabine will be administered at a dose of 10 mg/m2 subcutaneously (sc) twice daily (bid) from days 1-14. Triseonx will be administered at a dose of 0.25 mg/kg on days 1-5 and days 8-12. Trisenox will be restarted only when the QT interval returns to less than 500 msec. One treatment cycle consists of 2 weeks, with 14 days of cytarabine and 10 days of ATO.
  Subsequent cycles will be administered at the investigator's discretion, depending on response and tolerability. Patients may continue to receive treatment with Trisenox /LDAC for a period of up to 2 years as long as stable disease or clinical benefit and absence of unacceptable toxicity can be demonstrated.
Drug: cytarabine — Cytarabine will be administered at a dose of 10 mg/m2 subcutaneously (sc) twice daily (bid) from days 1-14. Trisenox will be administered at a dose of 0.25 mg/kg on days 1-5 and days 8-12. Trisenox will be restarted only when the QT interval returns to less than 500 msec. One treatment cycle consists of 2 weeks, with 14 days of cytarabine and 10 days of ATO.
  Subsequent cycles will be administered at the investigator's discretion, depending on response and tolerability. Patients may continue to receive treatment with Trisenox /LDAC for a period of up to 2 years as long as stable disease or clinical benefit and absence of unacceptable toxicity can be demonstrated.
  Other Names: cytosine arabinoside; Ara-C

SUMMARY:
This is an open-label, one arm, single institution study. Arsenic trioxide [TrisenoxTM Injection], 0.25mg/kg/dose administered intravenously over 2 hours.

20 patients

Complete remission, partial remission, clinical improvement, progressive disease, stable disease, relapse (per IWG consensus criteria, 2006) Clinical chemistry, hematology and ECGs will be assessed at least weekly during study treatments. Adverse events will be assessed in accordance with the NCI Common Toxicity Criteria, Version 2 at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > = 18 years with a documented history of myelofibrosis transformed to acute myeloid leukemia using the World Health Organization criteria of > = 20% blasts in the peripheral blood or bone marrow; the diagnosis of myelofibrosis could be either primary myelofibrosis (myelofibrosis with myeloid metaplasia, agnogenic myeloid metaplasia), post-polycythemia vera or post-essential thrombocytosis.
2. Patients > = 18 years with myelofibrosis (either primary (myelofibrosis with myeloid metaplasia, agnogenic myeloid metaplasia), post polycythemia vera or post essential thrombocytosis) who 1) meet the Mayo Clinic criteria for high risk disease (> = 2 of the following criteria: hemoglobin <10 g/dL, WBC <4 or >30 x 109/L, platelets < 100 x 109/L, absolute monocyte count > = 1 x 109/L) AND 2) have failed to respond to treatment with at least one prior therapy for myelofibrosis (erythropoietic cytokines, androgens, hydrea, interferon, thalidomide, lenalidomide or investigational therapy).
3. Patients must have discontinued prior myelofibrosis treatments (with the exception of hydrea, which is permitted for control of leukocytosis) for at least 14 days prior to starting study drug
4. ECOG performance status of < = 2
5. Serum creatinine < = 2.5 times the upper limit of normal
6. Serum bilirubin < = 2.5 times the upper limit of normal
7. Serum potassium >4.0 mEq/dL and serum magnesium >2.0 mg/dL. If these serum electrolytes are below the specified limits on the baseline laboratory tests, electrolytes will be administered to bring the serum concentrations to these levels before administering arsenic trioxide.
8. Patients will be eligible for this trial regardless of gender, racial/ethnic background, provided all other inclusion and exclusion criteria are met and the patient or patient's legally authorized guardian signs the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women
2. Presence of a (9;22) translocation cytogenetically, or presence of bcr-abl by FISH (fluorescence in situ hybridization) or PCR (polymerase chain reaction)
3. Absolute QT interval >500 msec in the presence of serum potassium ≥ 4.0 mEq/L and magnesium > = 1.8 mg/dL.
4. Prior cytotoxic chemotherapy for AML or MDS; prior treatment with hydroxyurea, 5-azacytidine, decitabine, thalidomide and lenalidomide are permitted. Prior treatment with low-dose cytarabine is not permitted.
5. Concurrent treatment with maintenance therapy, cytotoxic chemotherapy, radiation, or investigational agents.
6. Uncontrolled or severe cardiovascular, pulmonary or infectious disease or other medical condition that would prohibit use of the planned study treatments.
7. Inability or unwillingness to comply with the treatment protocol, follow-up, or research tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-02-08 (Actual)

PRIMARY OUTCOMES:
To assess the response rate in patients with advanced MF/LT using criteria of the International Working Group (IWG) | duration of study
To characterize the safety and tolerability of the regimen in this patient population | duration of study

SECONDARY OUTCOMES:
To assess overall survival | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Gail Roboz, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No